CLINICAL TRIAL: NCT06471140
Title: MRI Evaluation of Maternal Cardiovascular Response to Pregnancy in IVF Women Following Autologous Natural Cycle FET, Programmed FET and After Donor Embryo Transfer
Brief Title: Maternal Cardiovascular Adaption to Pregnancy in IVF Patients Following Frozen Embryo Transfer (FET)
Status: Enrolling by invitation | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: Regionshospitalet Viborg, Skive (Other)
Responsible Party: Principal Investigator, Lise Haaber Thomsen, MD, Consultant, Aalborg University Hospital
Other Study IDs: FET-PE-2024
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: IVF; Frozen Embryo Transfer (FET); Cardiovascular Adaption; Magnetic Resonance Imaging (MRI); Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IVF-pregnancy achieved following modified natural FET cycle, autologous embryo transfer: One corpus luteum, control group, autologous embryo transfer
  Interventions: Other: magnetic resonance imaging (MRI)
- IVF-pregnancy achieved following programmed FET cycle, autologous embryo transfer: No corpus luteum, study group, autologous embryo transfer
  Interventions: Other: magnetic resonance imaging (MRI)
- IVF-pregnancy achieved following egg donation in a FET cycle: One corpus luteum or no corpus luteum, study group, donor egg recipient.
  Interventions: Other: magnetic resonance imaging (MRI)

INTERVENTIONS:
Other: magnetic resonance imaging (MRI) — MRI performed three times during pregnancy and 6 months postpartum
  Other Names: Elastography; Seismocardiography

SUMMARY:
Aim of the study is to explore the effect of a lacking corpus luteum on maternal cardiovascular and metabolic adaption to pregnancy by the use of magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
The use of programmed frozen embryo transfer cycle (FET) in IVF women is associated with an increased risk of obstetric complications (pregnancy-induced hypertension, preeclampsia, postpartum hemorrhage and placenta accreta) compared to FET in natural cycle.

The lack of corpus luteum in programmed cycles and the subsequent absence of circulating vasoactive substances may lead to an impaired cardio-vascular adaption to pregnancy and thereby an increased risk of pregnancy-induced hypertension and preeclampsia.

The cardiovascular and metabolic adaption to pregnancy is evaluated throughout pregnancy by use of Magnetic Resonance Imaging (MRI) as well as non-invasive measurements by use of elastography and seismocardiography.

Patients are screened for preeclampsia throughout pregnancy with measurements of blood pressure, urine samples as well as blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Autologous embryo transfer in programmed FET-cycle or modified-natural FET-cycle or
* Planned donor egg transfer in programmed FET-cycle or modified-natural FET-cycle
* Age < 40 years
* BMI < 35
* Primary diagnosis being unexplained infertility, male infertility or tubal factor
* Singleton blastocyst transfer

Exclusion Criteria:

* PCOS
* Essential hypertension
* Diabetes Mellitus (type 1 or 2)
* Known cardiac disease
* Antiphospholipid syndrome, Lupus erythematosus, rheumatoid disease
* Preelampsia, gestational hypertension, gestational diabetes or severe intrauterine growth restriction (IUGR) in any previous pregnancy
* Smoking
* Multiple pregnancy
* Severe claustrophobia or any other contraindications to MRI

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: IVF-patients from The Fertility Unit Aalborg University Hospital and The Fertility Clinic, Skive Regional Hospital, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Maternal cardiovascular adaption to pregnancy | From early pregnancy to six months postpartum
Maternal metabolic adaption to pregnancy | From early pregnancy to six months postpartum
Placental function and fetal oxygenation estimated by longitudinal T2* weighted placental and fetal MRI | From early pregnancy to six months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Lise H Thomsen, MD, PhD, Study Chair — Department of Obstetrics and Gynecology, Aalborg University Hospital, Denmark; Anne N Sørensen, MD, PhD, Study Chair — Department of Obstetrics and Gynecology, Aalborg University Hospital, Denmark; Ulrik Kesmodel, Professor, Study Chair — The Fertility Unit, Department of Obstetrics and Gynecology, Aalborg University Hospital, Denmark; Peter Humaidan, Professor, Study Chair — The Fertility Clinic, Department of Obstetrics and Gynecology, Skive Region Hospital, Denmark
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark